CLINICAL TRIAL: NCT00290940
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Efficacy of CS-917 as Monotherapy for Type 2 Diabetes
Brief Title: Evaluation of Glucose Lowering Effect, Safety and Tolerability of CS-917
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS0917-A-U205
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Last update posted 2007-09-11 (Estimated); Status verified 2007-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes mellitus, Type 2; High blood sugar; Hyperglycemia; Antihyperglycemic agents; CS-917
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia | interventions — N,N'-((5-(2-amino-5-(2-methylpropyl)-4-thiazolyl)-2-furanyl)phosphinylidene)bis(alanine) diethyl ester; Metformin; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: CS-917
Drug: metformin hydrochloride
Drug: pioglitazone

SUMMARY:
This study will compare glucose lowering with CS-917 compared to placebo after 3 months of treatment

ELIGIBILITY:
Inclusion Criteria:

* Drug naive or newly diagnosed type 2 diabetic subjects:
* Never received oral antihyperglycemic or insulin therapy or
* No oral antihyperglycemic or insulin therapy for more than 6 months since original diagnosis and
* No insulin therapy within one year of screening, with the exception of use during hospitalization or for use in gestational diabetes and
* No antihyperglycemic therapy for more than three consecutive days, or a total of of seven non-consecutive days, during the 8 weeks prior to screening.
* HbA1C>6.7% and < or = to 10% at screening

Exclusion Criteria:

* Current insulin therapy
* Symptoms of poorly controlled diabetes
* History of diabetic ketoacidosis or hyperosmolar, nonketonic coma within one year of screening
* Serum bicarbonate < or = to 19 meq/L
* Serum creatinine (Scr) > 1.4 mg/dL (females) or 1.5 mg/dL (males)
* Contraindication to metformin

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2006-01; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in HbA1C after 12 weeks compared to placebo

SECONDARY OUTCOMES:
Onset of efficacy of CS-917
Safety and tolerability of CS-917
Changes in other relevant glycemic and metabolic measures
Proportion of subjects achieving therapeutic response
Proportion of subjects discontinuing or requiring rescue for continued or worsening hyperglycemia

CONTACTS AND LOCATIONS:
Locations (65):
- United States (65):
  - Birmingham, Alabama
  - Northport, Alabama
  - Mesa, Arizona
  - Phoenix, Arizona
  - Tempe, Arizona
  - Hot Springs, Arkansas
  - Cudahy, California
  - Long Beach, California
  - Roseville, California
  - Sacramento, California
  - Spring Valley, California
  - Studio City, California
  - Vista, California
  - Walnut Creek, California
  - West Hills, California
  - Wilmington, Delaware
  - Brooksville, Florida
  - Fort Lauderdale, Florida
  - Kissimmee, Florida
  - Miami, Florida
  - Pembroke Pines, Florida
  - Sebastian, Florida
  - St. Petersburg, Florida
  - Tallahassee, Florida
  - West Palm Beach, Florida
  - Rome, Georgia
  - Warner Robins, Georgia
  - Shawnee Mission, Kansas
  - Topeka, Kansas
  - Oxon Hill, Maryland
  - Cadillac, Michigan
  - Detroit, Michigan
  - Interlochen, Michigan
  - Livonia, Michigan
  - Port Gibson, Mississippi
  - Rolling Fork, Mississippi
  - Excelsior Springs, Missouri
  - Henderson, Nevada
  - Las Vegas, Nevada
  - Elizabeth, New Jersey
  - Toms River, New Jersey
  - Charlotte, North Carolina
  - Lenoir, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Delaware, Ohio
  - Marion, Ohio
  - Oklahoma City, Oklahoma
  - Beaver, Pennsylvania
  - Bensalem, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Reading, Pennsylvania
  - Anderson, South Carolina
  - Charleston, South Carolina
  - Greer, South Carolina
  - Nashville, Tennessee
  - Corpus Christi, Texas
  - Houston, Texas
  - Lake Jackson, Texas
  - North Richland Hills, Texas
  - San Antonio, Texas
  - Burke, Virginia
  - Olympia, Washington
  - Madison, Wisconsin